CLINICAL TRIAL: NCT05456399
Title: A Novel/Common Approach for Temporalis Muscle Thickness Measurement: Reliability and Agreement Study
Brief Title: A Novel/Common Approach for Temporalis Muscle Thickness Measurement
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğra İnce, Assoc. Prof, Bozyaka Training and Research Hospital
Other Study IDs: BITMA072022
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia; Stroke
MeSH Terms: conditions — Sarcopenia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cranial MRI: Axial sections of 5 mm thickness will be imaged. The thickness of the temporal muscle will be measured at the point where the floor of the temporal fossa is bounded most caudally by the zygomatic bone, sphenoid bone and temporal bone. After the MRI measurements are completed, the thickness of the muscle will be measured by ultrasound at the same location by two clinicians (a radiologist and a physiatrist) who are expertise in musculoskeletal ultrasonography.
- Patients with cranial CT: Axial sections of 5 mm thickness will be imaged. The thickness of the temporal muscle will be measured at the point where the floor of the temporal fossa is bounded most caudally by the zygomatic bone, sphenoid bone and temporal bone. After the MRI measurements are completed, the thickness of the muscle will be measured by ultrasound at the same location by two clinicians (a radiologist and a physiatrist) who are expertise in musculoskeletal ultrasonography.

SUMMARY:
The aim of this study is to propose a new measurement point for temporal muscle thickness (TMT) that can be similarly localized in computerized tomography (CT) /magnetic resonance imaging (MRI) and ultrasonography (USG), and to evaluate the reliability and consistency of these measurements.

DETAILED DESCRIPTION:
Recently, temporal muscle thickness (TMT) has been proposed as a new marker of whole-body muscle function. In addition, TMT has been shown to be a useful parameter for estimating skeletal muscle mass. Measurement of temporal muscle mass with CT and MRI has been studied in the literature in recent years. All stroke patients undergo cranial CT or MRI examinations at the time of admission. However, the literature indicates that USG can also be used to measure temporal muscle thickness. The recommended measurement points for CT, MRI, or USG in the studies performed to date depend on the particular imaging modality, and it does not seem possible to use them interchangeably. The aim of this study is to propose a new TMT measurement point that can be localized in a similar way in CT /MRI and USG, and to evaluate the reliability and agreement of these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Referral to the radiology department for an MRI or CT scan

Exclusion Criteria:

* Medically unstable condition (presence or high risk of impaired consciousness, respiration, or circulation).
* Vulnerable populations (patients with a terminal illness, people living in nursing homes, unemployed or poor people, people in need of urgent medical care, children, people unable to consent, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A tertiary health care facility
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Intra-rater reliability of ultrasonographic TMT measurement. | Baseline
  The intraclass correlation coefficient (ICC) of the two measurements performed by the physiatrist will be calculated using the "Two-way mixed effects, absolute agreement, single rater/measurement" model.
Inter-rater reliability of ultrasonographic TMT measurement. | Baseline
  Intraclass correlation coefficients of TMT measurements performed by the radiologist and physiatrist will be calculated using the "Two-way mixed effects, absolute agreement, multiple raters/measurements " model.
Inter-rater reliability of TMT measurements of MRI and CT | Baseline
  Intraclass correlation coefficients of TMT measurements performed by the radiologist and physiatrist will be calculated using the "Two-way mixed effects, absolute agreement, single rater/measurement " model.
Agreement of ultrasonographic TMT measurement with MRI and CT measurements. | Baseline
  The intraclass correlation coefficient of the measurements will be calculated using the "two-way mixed effects, absolute agreement, multiple raters/measurements" model. In addition, the agreement of the measurements will be evaluated using the Bland-Altman method. Furthermore, the Technical Error of Measurement (TEM) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Izmir Bozyaka Research and Education Hospital
Locations (1):
- Izmir Bozyaka Research and Training Hostpital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- [Background] Steindl A, Leitner J, Schwarz M, Nenning KH, Asenbaum U, Mayer S, Woitek R, Weber M, Schopf V, Berghoff AS, Berger T, Widhalm G, Prayer D, Preusser M, Furtner J. Sarcopenia in Neurological Patients: Standard Values for Temporal Muscle Thickness and Muscle Strength Evaluation. J Clin Med. 2020 Apr 28;9(5):1272. doi: 10.3390/jcm9051272. PMID 32354003
- [Background] Leitner J, Pelster S, Schopf V, Berghoff AS, Woitek R, Asenbaum U, Nenning KH, Widhalm G, Kiesel B, Gatterbauer B, Dieckmann K, Birner P, Prayer D, Preusser M, Furtner J. High correlation of temporal muscle thickness with lumbar skeletal muscle cross-sectional area in patients with brain metastases. PLoS One. 2018 Nov 29;13(11):e0207849. doi: 10.1371/journal.pone.0207849. eCollection 2018. PMID 30496307
- [Background] Katsuki M, Suzuki Y, Kunitoki K, Sato Y, Sasaki K, Mashiyama S, Matsuoka R, Allen E, Saimaru H, Sugawara R, Hotta A, Tominaga T. Temporal Muscle as an Indicator of Sarcopenia is Independently Associated with Hunt and Kosnik Grade on Admission and the Modified Rankin Scale Score at 6 Months of Patients with Subarachnoid Hemorrhage Treated by Endovascular Coiling. World Neurosurg. 2020 May;137:e526-e534. doi: 10.1016/j.wneu.2020.02.033. Epub 2020 Feb 14. PMID 32061954
- [Background] Nozoe M, Kubo H, Kanai M, Yamamoto M, Okakita M, Suzuki H, Shimada S, Mase K. Reliability and validity of measuring temporal muscle thickness as the evaluation of sarcopenia risk and the relationship with functional outcome in older patients with acute stroke. Clin Neurol Neurosurg. 2021 Feb;201:106444. doi: 10.1016/j.clineuro.2020.106444. Epub 2021 Jan 1. PMID 33395619